CLINICAL TRIAL: NCT00181051
Title: Clinical Utility of the Alaris MidLatencyAuditoryEvoked Potentials Monitor to Titrate the Anesthetic-Hypnotic Component of Anesthesia
Status: Suspended | Phase: Phase 3 | Type: Interventional
Sponsor: Gustave Roussy, Cancer Campus, Grand Paris (Other)
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PEA; CSET 2002/948
Record Dates: First submitted 2005-09-13; First posted 2005-09-16 (Estimated); Last update posted 2005-09-16 (Estimated); Status verified 2005-09

CONDITIONS: Scheduled General Anesthesia

INTERVENTIONS:
Device: Alaris AEP monitor

SUMMARY:
Index computed in real time from Auditory Evoked Potentials have been described parallel to depth of anesthesia. The goal of the study was to compare general anesthesia guided on Auditory Evoked Potentials monitoring to standrad practice in order to assess if AEP monitoring can improve recovery delay (main criteria) or intraoperative hemodynamic stability (secondary criteria). Patients were randomized in 2 groups, stratified by center. Group I : AEP guided anesthesia, Group II: Blind AEP record, standard practice.

ELIGIBILITY:
Inclusion Criteria:

* ASA status I-II patients
* aged 18 - 65 years
* scheduled for general surgery (except laparoscopic interventions) lasting longer than 1 hour.

Exclusion Criteria:

* Body weight < 70% or > 150% ideal body weight
* neurological disorder and hearing disorders (being not able to communicate with the patient in a normal tone)
* use of any medication interfering with pharmacological effect of the study including alcohol misuse or drugs.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 128
Dates: Start 2003-02

PRIMARY OUTCOMES:
Influence of AEP guided anesthesia on recovery delay

CONTACTS AND LOCATIONS:
Overall Officials: Michel STRUYS, MD, Principal Investigator — CHU de GENT - BELGIUM
Locations (1):
- Institut Gustave-Roussy, Villejuif, France